CLINICAL TRIAL: NCT05439278
Title: Randomized Phase III Study of Conventional Versus Hypofractionated Radiotherapy Combined With Temozolomide in Elderly Glioblastoma Patients
Brief Title: Conventional Versus Hypofractionated Radiotherapy With Temozolomide in Elderly Glioblastoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, Chan Woo Wee, M.D., Ph.D, M.D, PhD, Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KROG 21-11
Record Dates: First submitted 2022-06-21; First posted 2022-06-30 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Radiation Dose Hypofractionation; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypofractionated radiochemotherapy (Experimental): Radiotherapy: 40.05 Gy in 15 fractions (daily treatment, 5 per week) Temozolomide: concurrent (75 mg/m2/day qd) and adjuvant (6 cycles)
  Interventions: Radiation: Hypofractionated radiotherapy; Drug: Temozolomide
- Conventional radiochemotherapy (Experimental): Radiotherapy: 60 Gy in 30 fractions (daily treatment, 5 per week) Temozolomide: concurrent (75 mg/m2/day qd) and adjuvant (6 cycles)
  Interventions: Radiation: Conventional radiotherapy; Drug: Temozolomide

INTERVENTIONS:
Radiation: Hypofractionated radiotherapy — 40.05 Gy in 15 fractions (daily treatment, 5 per week)
  Arms: Hypofractionated radiochemotherapy
Radiation: Conventional radiotherapy — 60 Gy in 30 fractions (daily treatment, 5 per week)
  Arms: Conventional radiochemotherapy
Drug: Temozolomide — concurrent (75 mg/m2/day qd) and adjuvant (6 cycles)

SUMMARY:
In newly diagnosed glioblastoma patients aged 70 years or older who are suitable for concurrent temozolomide, the optimal dose of radiation therapy is controversial . The purpose of this study is to compare conventional radiotherapy of 60 Gy (6 weeks) versus hypofractionated radiotherapy of 40 Gy (3 weeks) in terms of overall survival as the primary endpoint along with progression-free survival, toxicity, quality of life, and prognostic biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed glioblastoma according to the 2021 World Health Organization classification
* interval of ≤4 weeks between pathological diagnosis and randomization
* aged 70 years or older
* gadolinium-enhanced MRI within 72 hours of surgery
* known o6-methylguanine-DNA-methyltransferase promoter methylation status
* Karnofsky performance score ≥60
* stable or decreasing dose of steroid (if necessary)
* no history of brain radiotherapy
* no history of any systemic chemotherapy
* adequate hematological, renal and hepatic functions for temozolomide
* able to start radiotherapy within 3 weeks from randomization

Exclusion Criteria:

* patients with spinal leptomeningeal carcinomatosis
* history of cancer other than the followings:
* carcinoma in situ of the cervix
* completely excised non-melanoma skin cancer
* cancers without any evidence of residual disease for 5 years or longer
* patients with serious active infection or other serious underlying medical conditions
* patients with psychological issues that cannot comply to the protocol
* patients with known hypersensitivity to temozolomide or compounds with similar chemical composition to temozolomide
* patients who are currently participating in other clinical trials

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | follow-up until 2 years
  from randomization

SECONDARY OUTCOMES:
progression-free survival | follow-up until 2 years
  from randomization
treatment-related toxicity | follow-up until 2 years
  any treatment-related toxicity
patient-reported quality of life | follow-up until 2 years
  European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30 version 3.0): range, 0-100 (a high score for a functional scale represents a high / healthy level of functioning; a high score for the global health status / QoL represents a high QoL; a high score for a symptom scale / item represents a high level of symptomatology / problems) Quality of Life Questionnaire-Brain Neoplasm (EORTC QLQ-BN20): range, 20-80; lower score means better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Chan Woo Wee, MD, PhD, Study Chair — Severance Hospital; In Ah Kim, MD, PhD, Study Chair — Seoul National University Bundang Hospital
Locations (1):
- Severance hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available.